CLINICAL TRIAL: NCT05067959
Title: Covid-19 Vaccine Responses in Patients With Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Shaare Zedek Medical Center (Other); Soroka University Medical Center (Other); Emek Medical Center (Other)
Responsible Party: Principal Investigator, IRIS DOTAN, Head of Gasteroenterology Division, Rabin Medical Center
Other Study IDs: 1072-20
Record Dates: First submitted 2021-06-21; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: IBD; Covid19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — complete blood count, CRP, Anti-TNF level and trough from relevant patients, COVID-19 serology including neutralizing antibodies, cytokine levels, lymphocyte subpopulation [CD4 CD8 B CD20/19, NKT], T cell proliferation, immunoglobulin levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients: patients with IBD (Chron's disease, Ulcerative colitis, IBD-Unspecify). patients will be divided into two sub-groups: IBD patients on anti-TNF therapy IBD patients on any other therapy
  Interventions: Biological: Covid-19 vaccine
- Controls: healthy volunteers
  Interventions: Biological: Covid-19 vaccine

INTERVENTIONS:
Biological: Covid-19 vaccine — blood tests and questioners before 1st vaccine, 3 weeks before 2nd vaccine, 4 weeks after 2nd vaccine, 6 months after 1st vaccine, and 12 months after 2nd vaccine

SUMMARY:
The 2019-coronavirus disease (COVID-19), caused by SARS-CoV-2, was identified as the source of pneumonia cases in Wuhan city in China. It rapidly spread worldwide and was declared by WHO as a pandemic. COVID-19 vaccines are expected to be the breakthrough in controlling the pandemic. However, studies performed only in healthy adults, and specifically excluded patients who were under immunomodulatory/biologic therapy, thus excluding patients with chronic inflammatory diseases (IBD). In this study we wish to understand vaccine efficacy and immunological response in IBD patients.

DETAILED DESCRIPTION:
Overall Aims:

1. To assess the immune response to COVID-19 vaccination in patients with IBD.
2. Comparing the short and long term immune response to vaccination among subgroups receiving different therapies.
3. To evaluate the different variables affecting immunity of these patients.
4. To assess adverse reactions to COVID-19 vaccines and IBD related complications.

Specifically:

1. To assess serologic response to COVID-19 vaccine(s) in patients with IBD treated with anti-TNF agents (+/- immunomodulators) compared to

   1. Healthy controls
   2. Patients with IBD not treated with anti-TNF (+/- immunomodulators)
2. To characterize serologic response: seroconversion, seroprotection and persistence of COVID-19 vaccine(s) in patients with IBD
3. To identify factors associated with serologic response
4. Side effects to vaccines
5. IBD exacerbation compared to activity at baseline
6. Symptomatic COVID-19

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults >18 years of age 2. Patients with either Crohn's disease, ulcerative colitis, ileostomy, pouch 3. Not vaccinated to COVID-19 [i.e. before 2 mRNA Pfizer vaccines provided, or before any vaccine provided as one injection 4. Ability to attend follow up visits 5. Ability to understand and sign an informed consent form

Exclusion Criteria:

* 1. Pregnant women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
vaccine efficacy in IBD population | 4 weeks post second COVID-19 vaccine.
  • Efficacy of the vaccination for IBD patients compared to the normal population measured as proportion of patients achieving positive serology

SECONDARY OUTCOMES:
Disease related variant affect immunological response | 12 months
  Measuring how the IBD disease activity (remission or flare) affect the response to the vaccine
Therapy related variants affect immunological response | 12 months
  Measuring how specific IBD therapies and doses, during induction or maintenance, interval between vaccination and anti TNF infusion/injection affect the response to the vaccine
Immunologic assessments affect response to vaccine | 12 months
  Measuring how immunoglobulin levels, lymphocyte subpopulations and HLA phenotype affect the response to the vaccine
Adverse Events to covid-19 vaccine | 12 months
  Following Adverse reactions to vaccines

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No